CLINICAL TRIAL: NCT06566248
Title: Randomized, Double-blind, Placebo-controlled Phase IIa Trial to Evaluate the Efficacy and Safety of Combined/Uncombined Nucleoside (Acid) Analogues of TQA3810 Tablets in Primary/Treated Patients With Chronic Hepatitis B
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of TQA3810 Tablets in Combination/Non Combination With Nucleoside (Acid) Analogues in Patients With Primary/Treated Chronic Hepatitis B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TQA3810-IIa-01
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: TQA3810 tablets+NUC (Experimental): Part A: TQA3810 tablets+NUC：A total of 4 dose groups were set up, which were respectively TQA3810 tablets 0.1mg once a day, 0.2mg once every two days, 0.3mg twice a week and 0.2mg once a day combined with oral nucleoside (acid) drugs (NUC) group for 24 weeks.
  Interventions: Drug: TQA3810 tablets+NUC
- Part A: Placebo+NUC (Placebo Comparator): Part A: Placebo+NUC: Placebo combined with oral nucleoside (acid) drugs (NUC) group was treated for 24 weeks.
  Interventions: Drug: Placebo+NUC

INTERVENTIONS:
Drug: TQA3810 tablets+NUC — TQA3810 is a novel, effective and highly selective small-molecule oral Toll-like receptors-8 agonist.
  Arms: Part A: TQA3810 tablets+NUC
Drug: Placebo+NUC — NUC:
  Entecavir Dispersible Tablets, Inhibit viral replication; Tenofovir Disoproxil Fumarate Tablets, Nucleotide reverse transcriptase inhibitors; Tenofovir Alafenamide Fumarate Tablets, Inhibit HBV replication.
  Arms: Part A: Placebo+NUC

SUMMARY:
To evaluate the efficacy and safety of combined/uncombined nucleoside (acid) analogues of TQA3810 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 (including boundary values), male or female.
* Serum virological criteria: serum HBsAg positive for more than 6 months or evidence of chronic hepatitis B for more than 6 months. During the screening period, 100 IU/ml≤HBsAg quantification ≤10000 IU/ml.
* No obvious cirrhosis was found by the researchers.
* The subjects can communicate well with the researchers, understand and comply with the requirements of this study, and understand and sign the informed consent.
* The 12-lead electrocardiogram was normal, or there were no clinically significant abnormal values as assessed by the investigator.

Treated patients must meet the following conditions:

* Subjects must have received oral nucleoside (acid) therapy (entecavir/ Tenofovir alafenamide Fumarate tablets/Tenofovir Disoproxil Fumarate Tablets) for ≥6 months prior to screening and stable treatment regimen for ≥3 months prior to screening.
* Patients with medical history 6 months or more before enrollment had HBV DNA< the lower limit of normal detection, and hepatitis B virus (HBV) DNA<20 IU/mL was detected by Roche COBAS Taqman during the screening period.

Newly treated patients need to meet the following conditions:

* At the time of screening, subjects had never received antiviral treatment for chronic hepatitis B (oral nucleoside drugs and interferon), or had received irregular antiviral treatment in the past, and had not received any antiviral treatment for chronic hepatitis B in the first 3 months of enrollment.
* HBV DNA≥2000 IU/mL(Roche COBAS Taqman).

Exclusion Criteria:

* Combined with other viral infections such as hepatitis A virus，hepatitis C virus, hepatitis D virus, hepatitis E virus, human immunodeficiency virus，syphilis (syphilis antibody positive by the researchers to determine the need for treatment). If hepatitis C virus (HCV) antibody positive, HCV RNA negative can not be excluded.
* Patients with significant fibrosis or cirrhosis before or at the time of screening: liver histopathological findings indicating Metavir F3 or F4 within 1 year before screening; FibroScan≥ 9.7 kPa 6 months before screening in treated patients and ≥ 12.4 kPa 6 months before screening in newly treated patients; Abdominal ultrasonography suggested suspected cirrhosis. Previous history of hepatic decompensation or screening period of hepatic decompensation, such as ascites, hepatic encephalopathy, esophageal and gastric varices bleeding, etc.
* Patients with a history of hepatocellular carcinoma (HCC) before or at the time of screening, or who may be at risk for HCC, such as suspicious nodules on imaging, or abnormal AFP (AFP>50ng/mL), should be excluded from HCC before enlisting.
* A history of malignant tumors within 5 years prior to screening, except for certain cancers that can be completely cured by surgical resection (such as skin basal cell carcinoma). Subjects being evaluated for active or suspected malignancy at the time of screening.
* Patients with other chronic liver diseases, including but not limited to autoimmune liver disease, alcoholic liver disease, hepatolenticular degeneration, etc.
* Have previously received organ transplantation and bone marrow transplantation.
* Patients with uncontrolled thyroid disease.
* Eye diseases: including fundus lesions (cotton wool changes in the fundus with symptoms) and retinopathy.
* Autoimmune diseases include but are not limited to: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, sarcoidosis, psoriasis, autoimmune uveitis, etc.
* Current alcohol and drug abuse was determined by the investigator. Subjects with a history of excessive alcohol use. A history of excessive alcohol use was defined as alcohol consumption >210g per week for men and >140g for women in the past 12 months. Alcohol intake (g) = amount of alcohol consumed (ml) × alcohol degree % × 0.8.
* Blood transfusion ≤2 months before screening and/or blood donation ≤1 month before screening. Note: Subjects were not allowed to donate blood throughout the study period.
* Have a history of allergy to the experimental drug or its excipients;
* Female subjects are pregnant, breastfeeding or have positive pregnancy results during the screening period or during the test;
* Those that researchers believe should not be included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) during the study period | Up to 52 months
  The study required collection of any adverse medical events, whether causally associated with the investigational drug or not, from the time the subject signed the informed consent to 28 days after the end of study medication or the initiation of other anti-HBV therapy (whichever came first).

SECONDARY OUTCOMES:
Changes in serum HBsAg | 24 weeks
  Changes in serum HBsAg from baseline at 24 weeks
HBV DNA level changes and drug resistance monitoring | 24 weeks
  Changes in HBV DNA levels from baseline and drug resistance monitoring.
HBeAg level change | 24 weeks
  Changes in HBeAg levels from baseline.
HBsAg clearance and/or serological conversion | 24 weeks
  Percentage of subjects with HBsAg clearance and/or serological conversion.
HBeAg clearance and/or serological conversion | 24 weeks
  Percentage of subjects with HBeAg clearance and/or serological conversion
HBsAg level decreased by ≥0.5log10 IU/ml | 24 weeks
  Proportion of subjects with HBsAg levels decreased at least 0.5log10 IU/ml
Changes of HBV RNA and hepatitis B core-related antigen (HBcrAg) levels during treatment | 24 weeks
  Changes of HBV RNA and HBcrAg levels from baseline during treatment
Peak time (Tmax) | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  Time to peak blood concentration after a single dose.
Peak Concentration | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The highest plasma drug concentration that can be achieved after medication.
Area under blood concentration-time curve (AUC) | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The amount of drug absorbed into the human circulation after a single dose can be estimated using the area under the blood concentration-time curve.
Apparent volume of distribution (Vd/F) | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  When a drug reaches homeostasis in the body, the ratio of the amount of drug in the body to the blood concentration is called the apparent volume of distribution.
Plasma clearance | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  How many milliliters of plasma can the kidneys completely clear in unit time (per minute).
Elimination half-life time | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The time it takes for the plasma concentration to drop by half
Peaking Time | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The time required to reach peak steady-state concentration after administration.
Steady state maximum concentration | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The highest blood concentration that occurs After stabilization
Steady state minimal concentration | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The lowest blood concentration that occurs after stabilization.
Area under steady-state blood concentration-time curve | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  The area under the curve obtained with blood drug concentration as the vertical axis and time as the horizontal axis after administration.
Evaluate whether TQA3810 will affect the heart rate-corrected QT interval (QTc) of newly treated/treated chronic hepatitis B patients | 24 weeks
  Evaluate whether TQA3810 will affect the QTc interval of newly treated/treated chronic hepatitis B patients
Pharmacodynamic characteristics (IFN-γ, IL-1RA, CCL2, CCL4, CCL8, CCL11, CCL20, CXCL8, IL-12p70, IL-12p40, TNF-α, CRP) | In 60 minutes pre-dose on day 1, 0.5, 1, 2, 4, 12 hours after dose; Day 15 within 60 minutes pre-dose; Day 29 within 60 minutes pre-dose; Day 57 within 60 minutes pre-dose; Day 85 within 60 minutes pre-dose, 0.5, 1, 2, 4, 12 hours after dose
  Characteristics of IFN-γ, interleukin-1 receptor antagonist (IL-1RA), chemokine (C-C motif) ligand 2 (CCL2), Chemokine (C-C motif) ligands 4 (CCL4) , Chemokine (C-C motif) ligands 8 (CCL8), Chemokine (C-C motif) ligands 11 (CCL11), Chemokine (C-C motif) ligands 20 (CCL20), C-X-C motif chemokine ligand 8 (CXCL8), IL-12p70, IL-12p40, Tumor necrosis factor-α (TNF-α), C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Zunyi Medical University Affiliated Hospital, Zunyi, Guizhou
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - Shenyang Sixth People's Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi